CLINICAL TRIAL: NCT00180011
Title: Efficacy of Omalizumab as Add on Therapy for Minority Patients With Moderate to Severe Asthma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: DiMango, Emily, M.D. (Individual)
Collaborators: Genentech, Inc. (Industry); Novartis (Industry)
Responsible Party: Principal Investigator, Emily DiMango, Assistant Professor, DiMango, Emily, M.D.
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 20041332
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Asthma
Keywords: omalizumab; severe asthma; moderate asthma; injectable asthma medication; Xolair
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- omaluzimab (Experimental)
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Omalizumab — injectable medication

SUMMARY:
This study will be a randomized, placebo controlled, double blind study to measure the safety and efficacy of a new, injectable asthma medication, omalizumab, in a group of minority with moderate to severe asthma who are not adequately controlled with use of inhaled or oral steroids. Primary endpont will be change in asthma symptom utility index. Secondary endpoints will be changes in asthma Quality of life, asthma exacerbation rate, and lung function over the 12 week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30
* Minority Patients
* Moderate or Severe allergic asthma (as defined by the National Asthma Education and Prevention Guidelines(7)]. Allergic asthma will be defined as elevated IgE level (> 100 IU/ml) and skin test sensitivity to at least one common aeroallergen
* asthma control score greater than 1.5 (5) at randomization visit with use of equivalent of at least 1000 mcg fluticasone daily or systemic steroid use
* FEV1 50-90% predicted at screening and randomization visit

Exclusion Criteria:

* Active smoking within one year and/or greater than 10-pack year history of smoking
* Women of childbearing age must be using effective contraception
* Malignancy diagnosed within the past 5 years
* Underlying lung disease other than asthma
* Inability to comply with study protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2005-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Asthma symptom utility index | 6 months

SECONDARY OUTCOMES:
Secondary endpoints will be changes in asthma Quality of Life, asthma exacerbation rate, and lung function over the 12 week treatmet period. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Emily DiMango, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States